CLINICAL TRIAL: NCT05262075
Title: Experiences of an Online Mindfulness Program Integrating Resiliency Factors for Women Who Have Experienced Intimate Partner Violence
Brief Title: Online Mindful & Resiliency Program Intimate Partner Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Dragana Krpalek, Associate Professor, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5210387
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Mindfulness; Intimate Partner Violence
Keywords: Mindfulness; Resiliency; Online; Domestic violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness and Resiliency Program (Experimental): This is an online mindfulness program that integrates resiliency factors to women
  Interventions: Other: Online Mindfulness Resiliency Program

INTERVENTIONS:
Other: Online Mindfulness Resiliency Program — An approximate 20 minute online mindfulness resiliency program offered 3/wk x 4 weeks.

SUMMARY:
The purpose of this study is to explore the experiences and benefits of offering an online mindfulness program that integrates resiliency factors to women.

DETAILED DESCRIPTION:
The purpose of this study is to explore the experiences and benefits of offering an online mindfulness program that integrates resiliency factors to women. Investigators will recruit participants via email and social media flyers to local community sites as well as approved Loma Linda University affiliated sites. Participants who consent will then complete a Demographic Questionnaire(before initial session of program), Pre and Post Stress Surveys (at the start and end of each session), Five-Facet Mindfulness Questionnaire(before and after completion of the program), and a semi-structured interview after the completion of the program. The program will be done be 20-minutes sessions for 3x/week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women who self-identify as having or who are currently experiencing intimate partner violence
* English or Spanish speaking
* Between 18 and 85 years old.

Exclusion Criteria:

* Males
* No experience of partner violence
* Not fluent in either English or Spanish <18 and >85 years of age

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Level of Stress | Change between Baseline and Week 5 of mindfulness training
  Participants rate their stress level at the beginning and end of each session on a scale of 1-10.
Level of Self-Awareness | Change between Baseline and Week 5 of mindfulness training
  Self-reported 15-item questionnaire designed to provide information on self-awareness and suggests how effective mindfulness practices are. Responses will be recorded on a Likert scale from 0 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Dragrana Krpalek, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No